CLINICAL TRIAL: NCT05203094
Title: Urdu Version of Tinetti Balance and Gait Assessment Scale, (Performance-oriented Mobility Assessment) Reliability and Validity Study
Brief Title: Urdu Version of Tinetti Balance and Gait Assessment Scale,(POMA),Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00281
Record Dates: First submitted 2022-01-08; First posted 2022-01-24 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Balance; Distorted
Keywords: Assessment,balance ,older people, reliability,validity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study we will observe the reliability and validity of Tinetti Balance assessment scale,(POMA) in Urdu language in Pakistani geriatric population with balance impairment. Also, check the improvement in assessment and rehabilitation in geriatrics with balance problem.

DETAILED DESCRIPTION:
The aim of study is to translate and culturally adapt Tinetti balance assessment scale (POMA) into Urdu language and secondly to investigate the reliability and validity of Tinetti Balance assessment scale (POMA) in geriatrics Pakistani population.This study will be cross sectional survey study in which convenience sampling technique will be used. Two scales will be performed by patient Tinetti Balance assessment scale and Berg Balance Scale (evaluate balance), Timed Up and Go Test (TUGT) (measure functional mobility) for comparison and data will be collected. The results of study will help to know the validity and reliability of Tinetti Balance assessment scale (POMA) in Urdu version with balance impairments in geriatric population.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk a minimum of 6m with or without a walking Aid
* observed balance impairment evaluated subjectively by a physical therapist during the initial training session (Berg Balance scale and time up and go test )

Exclusion Criteria:

* people with amputated lower extremities using prosthetic leg
* those who underwent orthopedic surgery within the last 6 weeks
* Dependent on wheel chairs and bed ridden patients
* Dementia and Alzheimer's patients
* illiterate people

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: older people,especially age-related impairments in balance and postural control that effect the performance of everyday activities, which are primary reasons for falls. about 28-35% of older people (65 years) are experiencing falls. the prevalence increases to 50%up to 80 years of age
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Tinetti balance and gait assessment scale (POMA) | 1st day
  tinetti balance and gait assessment scale is used to evaluate older people's ability to maintain postural balance and gait, it is composed of two separate categories as balance and gait test balance and gait are evaluated with nine and eight items, respectively. the total score of scale 28 points. the highest score indicates the best performance
Tinetti balance and gait assessment scale (POMA) | 2nd day
  tinetti balance and gait assessment scale is used to evaluate older people's ability to maintain postural balance and gait, it is composed of two separate categories as balance and gait test balance and gait are evaluated with nine and eight items, respectively. the total score of scale 28 points. the highest score indicates the best performance

SECONDARY OUTCOMES:
berg balance scale | 1st day
  the berg balance scale is an objective assessment of balance performance based on 14 items common to daily activities. it is a 14 items scale that rate 0 (unable to perform) to 4 (normal performance) for each item. the total score is 56 points, high score higher balance ability

OTHER OUTCOMES:
Timed Up and Go Test | 1st day
  screening test that is measure functional mobility in older adults

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No